CLINICAL TRIAL: NCT06523283
Title: The Effect of the Use of Natural Landscape Pictures Accompanied by Music on Breastfeeding, Breastfeeding Satisfaction and Maternal Attachment to Lactation-Period Mothers During Breastfeeding
Brief Title: The Effect of Nature Images Accompanied by Music on Breastfeeding, Breastfeeding Satisfaction and Maternal Attachment"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, NURAY AYDIN, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HasanKU-SBF-RK-01
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Breast Feeding
Keywords: Breast Feeding; Maternal attachment; Music therapy; Maternal Satisfaction
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: One intervention group and one control group
Who Masked: Outcomes Assessor
Masking Description: outcome assesments will be performed by statistician who has blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Landscape Pictures Accompanied by Music İntervention Group (Experimental): Natural Landscape Pictures Accompanied by Music video will be applied to interevention group. They will watch the video for 10 sessions.
  Interventions: Other: Natural Landscape Pictures Accompanied by Music
- Control group with no intervention (No Intervention): Control group will not receive any intervention.

INTERVENTIONS:
Other: Natural Landscape Pictures Accompanied by Music — after data collection tools filled by participants , they will watch the video one time in hospital bed while breastfeeding , second time in their home while researchers is there and they will also receive the video link so they will contunie to watch video 8 more time. in total 10 sessions will be completed.
  Arms: Natural Landscape Pictures Accompanied by Music İntervention Group

SUMMARY:
The study was planned as a randomized controlled study to evaluate the effect of using natural landscape pictures accompanied by music during breastfeeding for lactating mothers on breastfeeding, breastfeeding satisfaction and maternal attachment.

DETAILED DESCRIPTION:
This research is planned as a randomized controlled study to evaluate the effect of using natural landscape pictures accompanied by music during breastfeeding on breastfeeding, breastfeeding satisfaction, and maternal attachment in lactating mothers.

The research will be conducted with primiparous mothers who apply to Adıyaman University Training and Research Hospital Gynecology clinics between January 2024 and August 2024 and meet the inclusion criteria. The study will include a total of 90 participants, divided into one intervention group and one control group.

As a pre-test, the Socio-Demographic Data Survey, LATCH Breastfeeding Diagnosis and Evaluation Scale, Visual Analogue Scale for Satisfaction Evaluation, and Maternal Attachment Scale will be administered to mothers who have just given birth at the clinic. Both groups will receive breastfeeding education.

For the intervention group, mothers will watch nature scene pictures accompanied by music prepared by the researcher. This will be done once in the hospital, once during a home visit after discharge, and then daily at home, with the researcher checking in by phone to ensure the mothers watch the scenes eight more times. The intervention will be conducted a total of 10 times.

Finally, the data collection phase will be completed by administering the post-test surveys to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreeing to participate in the research
* Being over 18 years old
* Being at least a primary school graduate
* Not having a diagnosed psychiatric disease
* Without mental disability
* Turkish speakers and those who do not have communication problems
* Primiparous mothers
* The mother does not have any problems that would prevent her from breastfeeding (e.g., nipple cracks)
* The child is not premature
* Mothers who gave birth at term
* The baby is not low birth weight
* Mothers who do not have any problems that would prevent the baby from breastfeeding

Exclusion Criteria:

* Being illiterate
* Being under 18 years old
* Having a diagnosed psychiatric illness
* Having mental disability and communication problems
* Those who do not speak Turkish and have communication problems
* Non-primiparous mothers
* The mother has any problems that may prevent her from breastfeeding (e.g., nipple cracks)
* Having a premature baby
* Mothers who did not give birth at term
* Low birth weight of the baby
* Mothers who have any problems that may prevent the baby from breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-08-02 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Socio-Demographic Data Survey | Ten days
  It consists of 14 questions about the sociodemographic characteristics of mothers, prepared by the researcher through a literature review on the subject and in line with the suggestions of the thesis monitoring committee members."
LATCH Breastfeeding Diagnostic and Evaluation Scale | Ten days
  It is a diagnostic method used to evaluate breastfeeding success, first created in 1986 by likening it to the APGAR score system in terms of scoring method. The average application time varies between 7-10 minutes. It consists of five evaluation criteria, and the abbreviation of the first letters of the English equivalents of these criteria forms the name of the scale. L; latch on the breast, A; audible swallowing, T; type of the nipple, C; comfort breast/nipple, and H; hold/help. Each item is evaluated between 0-2 points. The highest total score that can be obtained is 10, and a high score indicates high breastfeeding success. The Turkish reliability study of the tool was conducted by Yenal and Okumuş, and it was found to be a suitable and reliable diagnostic tool for use. While the Cronbach's alpha value of the original form of the scale was found to be 0.93, it was found to be 0.95 in the Turkish adaptation study.
The Visual Analog Scale (VAS) | Ten days
  It is an extremely simple, effective, and repeatable measurement tool that requires minimal equipment and can be used to measure pain, nausea, vomiting, and satisfaction. The VAS is a 10 cm long scale drawn horizontally or vertically. The easiest way to assess satisfaction is to ask the individual if they are satisfied. However, a yes or no answer is not sufficient to evaluate satisfaction. Therefore, the use of a scale in assessing satisfaction transforms the quality of satisfaction described by individuals/patients with numbers or words into an objective measure, eliminating different interpretations among the healthcare team providing patient care. The visual analog scale consists of numbers ranging from 0 to 10. In evaluating patient satisfaction, 0 is considered not at all satisfied and 10 is considered very satisfied.
Maternal Attachment Scale | Ten days
  Each item is a 26-item, four-point Likert scale ranging from "always" to "never." Each item contains direct statements and is scored as follows: Always (a) = 4 points, Often (b) = 3 points, Sometimes © = 2 points, and Never (d) = 1 point. A high score indicates a high level of maternal attachment. The lowest score obtainable from the scale is 26, and the highest score is 104.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray Aydın, Master, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Adiyaman University Education and Research Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No